CLINICAL TRIAL: NCT01577004
Title: Do Apolipoprotein E Polymorphisms Influence Risk of Cognitive Decline by Modulating Omega-3 Fatty Acid Metabolism?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, Assistant Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AFMNet-1; Discovery grant (Other Grant/Funding Number: Advanced Foods and Materials Network)
Record Dates: First submitted 2012-02-24; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omega-3 fatty acid supplement (Experimental): Data obtained after the intervention was compared to baseline data
  Interventions: Dietary Supplement: omega-3 fatty acid

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — Subjects will be given four 1 g capsules of fish oil providing 1.4 g/d of EPA and 1.0 g/d of DHA as ethyl esters (Ocean Nutrition, Dartmouth, NS), which is similar to the dose used in previous studies with MCI and AD (20, 21).
  Other Names: Ocean Nutrition, Dartmouth, NS

SUMMARY:
BACKGROUND: Compared to the epsilon 2 or epsilon 3 alleles, the epsilon 4 allele of apolipoprotein E (ApoE4) is associated with twice the prevalence of late-onset Alzheimer's disease (AD). Epidemiological studies show that risk of AD varies inversely with consumption of omega-3 fatty acids from fish and seafood. Despite apparently lower fish intake in AD, pooled analysis of the literature shows that plasma and brain docosahexaenoic acid (DHA) is actually the same in AD as in healthy age-matched controls. Fish oil trials in AD are also not convincing. We recently shown that ApoE4 carriers have 41% higher fasting plasma EPA and DHA compared to non-carriers, but the plasma EPA and DHA response to fish oil in ApoE4 carriers was half that seen in non-carriers.

HYPOTHESES: (i) Carriers of ApoE4 have altered metabolism of carbon-13 (13C)-DHA as well as EPA and DHA provided in a dietary supplement. (ii) A dietary supplement of EPA+DHA will improve cognitive performance but only in non-carriers of ApoE4.

OBJECTIVES: In both carriers and non-carriers of ApoE4, to compare whether- i) ApoE4 alters incorporation of 13C-DHA into plasma lipids or its beta-oxidation.

ii) 13C-DHA metabolism changes while on a dietary supplement of EPA+DHA; iii) Better cognitive performance occurs while on EPA+DHA and is linked to raising plasma EPA and/or DHA.

EXPERIMENTAL METHODS: Participants older than 50 y old and not demented were enrolled. DHA metabolism was evaluated using both 13C-DHA and an EPA+DHA supplement (2.4 g/d for 5 mo; n = 20/gp). Before and in the last month of supplementation, plasma uptake and beta-oxidation of 50 mg of 13C-DHA was followed during one month. Blood omega-3 fatty acids was evaluated monthly during the supplementation period. Cognitive testing was performed before and 4 months after starting the omega-3 fatty acid supplement.

IMPLICATIONS: This project will help explain the apparent link that is newly emerging between ApoE polymorphisms, altered omega-3 fatty acid metabolism and risk of cognitive decline, and should help in the development of nutraceutical-based clinical trials using fish oil for the elderly.

DETAILED DESCRIPTION:
To come

ELIGIBILITY:
Inclusion Criteria:

* MCI will be defined by Winblad et al. (33), with diagnosis confirmed by a geriatrician through neuropsychological evaluation done within the last 6 months.
* if diagnosis was done more than 6 months ago, the subject will be re-evaluated before inclusion to confirm MCI rather than conversion to AD.

Exclusion Criteria:

* tobacco
* malnutrition (assessed from blood albumin, haemoglobin and lipids)
* subjects already taking an EPA+DHA supplements
* swallowing problems, uncontrolled diabetes (raised fasting glucose, haemoglobin A1c)
* uncontrolled thyroid disease
* severe renal failure
* chronic immune condition or inflammation (raised C-reactive protein, white cell count)
* cancer
* recent major surgery or cardiac event
* uncorrected visual or hearing problems
* dementia
* ongoing or past severe drug or alcohol abuse
* psychiatric difficulties or depression as evaluated by the geriatric depression scale test (34)
* use of psychotropic medications except for short-acting benzodiazepines taken before sleep.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
13C-DHA incorporation into plasma lipids or beta-oxidation. | one month
  Before and in the last month of supplementation, plasma incorporation and beta-oxidation of 50 mg of 13C-DHA will be followed during one month. Blood and breath samples will be collected at time 0 h, 1 h, 2 h, 4 h, 6 h, 8 h, 24 h, 7 d, 14 d, 21 d, and 28 d.

SECONDARY OUTCOMES:
Cognitive performance compared to baseline | 5 month
  Cognitive testing was done before and 4 months after starting the omega-3 fatty acid supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Plourde, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Melanie Plourde, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Plourde M, Chouinard-Watkins R, Rioux-Perreault C, Fortier M, Dang MT, Allard MJ, Tremblay-Mercier J, Zhang Y, Lawrence P, Vohl MC, Perron P, Lorrain D, Brenna JT, Cunnane SC. Kinetics of 13C-DHA before and during fish-oil supplementation in healthy older individuals. Am J Clin Nutr. 2014 Jul;100(1):105-12. doi: 10.3945/ajcn.113.074708. Epub 2014 May 14. PMID 24829492